CLINICAL TRIAL: NCT00702962
Title: Phase I/II Study of Carboplatin and Etoposide in Combination With Vorinostat for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Carboplatin and Etoposide in Combination With Vorinostat for Patients With Extensive Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Chandra P. Belani, Professor of Medicine, Milton S. Hershey Medical Center
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSHCI 08-005
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-09

CONDITIONS: Small Cell Lung Cancer
Keywords: lung cancer; small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Vorinostat; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I: Vorinostat 200 mg (Experimental): Vorinostat 200 mg PO QD D1-14; Administer with Carbo 6 (AUC) D3; Etoposide 100 mg/m2 D1,2,3 "Vorinostat", "Carboplatin", "Etoposide"
  Interventions: Drug: Vorinostat, Carboplatin, Etoposide

INTERVENTIONS:
Drug: Vorinostat, Carboplatin, Etoposide — Study originally a Phase I standard dose escalation of the study medication Vorinostat with sequential cohorts of 3-6 participants entered to 3 dose levels (200mg, 300mg, 400mg). Dose escalation stopped after participant 1 on dose level 2 due to recently published research identifying an appropriate dosing regimen. A set dose was then to be administered to all subsequent participants. This regimen (a "cycle") consisted of Vorinostat on Day 1 through Day 4, Carboplatin AUC 6 on Day 3, and Etoposide 100 mg/m2 on Day 3 through Day 5. Treatment cycles were repeated every 21 days (3 weeks) for 4 cycles total.
  Other Names: Suberoyl anilide hydroxamic acid (SAHA)

SUMMARY:
The Phase I portion of the study is to assess the maximum tolerated dose of vorinostat when combined with carboplatin plus etoposide. The Phase II portion is to determine progression-free survival among patients with extensive disease small cell lung cancer receiving carboplatin plus etoposide with vorinostat.

DETAILED DESCRIPTION:
Vorinostat inhibits growth and induces apoptosis in various human carcinoma cells. Furthermore, it affects the expression of various genes that are necessary for proliferation of cancer cells. Vorinostat also appears to block angiogenic signaling. Pre-treating four human cancer cell lines (including a brain tumor line) with vorinostat increased the killing efficiency of etoposide, ellipticine, doxorubicin, or cisplatin, but not of the topoisomerase I inhibitor camptothecin 13. Topoisomerase II is a ubiquitous nuclear enzyme that is involved in DNA replication, transcription, chromosome segregation, and apoptosis. It is the target for several anti-cancer drugs including etoposide. Treatment with HDAC inhibitors induces expression of topoisomerase II in cancer cells and enhances the sensitivity to etoposide 14.

Early phase clinical trials have demonstrated single agent anti-cancer activity with vorinostat. In our study, combination of vorinostat with carboplatin and paclitaxel, demonstrated promising anticancer activity against NSCLC, including histological subsets of patients whose tumors demonstrated neuroendocrine differentiation 8. For all these reasons, vorinostat is a rational choice to combine with the regimen of carboplatin and etoposide for evaluation in patients with SCLC-ED.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with CT scan.
* Patients must be chemotherapy naive.
* Previous radiotherapy is allowed only if < 30% of marrow bearing bones were irradiated and if radiotherapy was completed at least 2 weeks prior to enrollment and the patient has recovered from all adverse effects of prior radiotherapy.
* Age >18 years.
* Life expectancy of greater than 3 months.
* ECOG performance status <2 (Karnofsky >60%).
* Adequate organ and marrow function.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or double barrier method of birth control) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have had chemotherapy or any other investigational agent for any indication within 30 days of study enrollment.
* Patients who have had radiotherapy within 2 weeks, prior to entering the study or those who have not recovered from adverse events due to these therapies.
* Patients with known brain metastases are excluded.
* Patients who have been previously treated with an HDAC inhibitor (use of valproic acid is allowed with a 30-day washout).
* Patients with peripheral neuropathy CTC grade >2 are excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any major surgery within 2 weeks prior to enrollment. Minimally invasive procedures for the purpose of diagnosis or staging of the disease are permitted.
* History of another malignancy in the last 5 years. Patients with prior history of in situ cancer, basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone and have been continuously disease free for at least 5 years.
* Pregnant women are excluded from this study because irinotecan and paclitaxel are antineoplastic agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with agents used in this trial, breastfeeding should be discontinued if the mother is treated with these agents.
* Patients with known HIV, Hepatitis B, Hepatitis C or active Hepatitis A are excluded.
* Patients on any systemic steroids for any indication, with doses that have not been stabilized to the equivalent of < 10 mg/day prednisone during the 30 days prior to study enrollment. This does not include short courses of steroids administered at high doses.
* Patients with the inability to absorb oral vorinostat.
* Patients with known allergy or hypersensitivity to any component of any of the study therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P Belani, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
To determine if data is valuable

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open to accrual 09/2008 as Phase I study. Three participants treated with dose level 1. Similar NCI-CTEP Phase I trial (NCI 8703) established the maximum tolerated dose (MTD) for the study drug. This study was amended to Phase II using the NCI established dose. One participant treated on Phase II. Closed to accrual 01/2012 due to low enrollment.
Pre-assignment Details: Eight patients total were consented (i.e. "enrolled"). Three of the 8 were determined to be ineligible upon screening. One of the 8 was eligible but subsequently declined participation soon after signing consent. Four (4) of 8 enrolled went to active treatment ("started"). Of these 4, 3 participated in Phase I and 1 participated in Phase II.
Groups:
- Phase II Portion - Vorinostat 300mg: Phase 2 is to determine progression free survival among patients with extensive disease SCLC receiving carboplatin plus etoposide with vorinostat.Vorinostat, Carboplatin, Etoposide, SAHA
  SAHA: Once the recommended phase II dose has been established and additional 15 patients will be enrolled. Days 1-4 Vorinostat recommended phase II dose po QD;Day 3 Carboplatin 6 AUC; Days 1,2,3 Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each patient. An additional 35 patients on the phase II portion of the trial will be required to achieve the outlined objectives.
- Phase I Portion - Vorinostat 200mg: Vorinostat 200 mg PO QD D1-14; Carbo 6 (AUC) D3; Etoposide 100 mg/m2 D1,2,3 Vorinostat, Carboplatin, Etoposide, SAHA.
  Vorinostat, Carboplatin, Etoposide: Sequential cohorts of 3-6 patients will be entered to the following dose levels: Level 1 - Days 1-14: Vorinostat 200 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Level 2 - Days 1-14: Vorinostat 300 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2; Level 3: Days 1-14: Vorinostat 400 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each patient. Phase I was prematurely closed as an NCI study established the MTD. This study proceeded to Phase II soon after the first participant was enrolled at Dose Level 2 (300mg).
Period: Overall Study
Arm/Group | Phase II Portion - Vorinostat 300mg | Phase I Portion - Vorinostat 200mg
Started | 1 (One initiated treatment. Milestones not achieved due to premature closing due to low accrual.) | 3 (Three treated. Milestone not met as Phase I closed prematurely as NCI research established the MTD.)
Completed | 0 (The one participant off treatment after 2 doses due to concurrent health disorder.) | 2 (Two completed all required cycles. One experienced progressive disease after 2 cycles)
Not Completed | 1 | 1
Not completed — Progressive disease | 0 | 1
Not completed — Hospitalized for other health disorder | 1 | 0

BASELINE CHARACTERISTICS:
Population: The first Phase I portion enrolled the first 3 participants at dose level 1 (Vorinostat 200 mg). Phase I closed prematurely as the recommended dose was established in other national clinical trials. Phase II used the established dose of Vorinostat 300 mg. Phase II closed prematurely due to low accrual.
Groups:
- PHASE I: Vorinostat 200mg Carbo 6 (AUC): Phase I portion: To determine MTD of Vorinostat when used in combination with other chemotherapy. Start at Vorinostat 200 mg PO QD D1-14; Carbo 6 (AUC) D3; Etoposide 100 mg/m2 D1,2,3; Vorinostat, Carboplatin, Etoposide, SAHA
  Vorinostat, Carboplatin, Etoposide: Sequential cohorts of 3-6 patients will be entered to the following dose levels: Level 1 - Days 1-14: Vorinostat 200 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Level 2 - Days 1-14: Vorinostat 300 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2; Level 3: Days 1-14: Vorinostat 400 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each patient.
- PHASE II: Vorinostat 300mg Carbo 6 (AUC): Phase II portion: To determine progression free survival among patients with extensive disease SCLC receiving carboplatin plus etoposide with fixed dose Vorinostat. (Vorinostat, Carboplatin, Etoposide, SAHA)
  SAHA: Once the recommended phase II dose has been established and additional 15 patients will be enrolled. Days 1-4 Vorinostat recommended phase II dose po QD;Day 3 Carboplatin 6 AUC; Days 1,2,3 Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each patient. An additional 35 patients on the phase II portion of the trial will be required to achieve the outlined objectives.
- Total: Total of all reporting groups
Arm/Group | PHASE I: Vorinostat 200mg Carbo 6 (AUC) | PHASE II: Vorinostat 300mg Carbo 6 (AUC) | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.8) | 70 (0) | 65.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Assess Maximum Tolerated Dose of Vorinostat When Combined With Carboplatin and Etoposide of Patients With Extensive Disease SCLC
Description: To estimate the maximum tolerated dose of vorinostat using a traditional dose escalation schedule ("3 + 3 design). MTD is determined by assessing for specific predefined dose limiting toxicities. A starting dose of vorinostat 200mg was combined with carboplatin and etoposide. Dose escalation went in increments of 100mg (i.e. 300mg, 400mg).
Time Frame: 2 years, not analyzed
Population: The first three participants enrolled were treated at dose level 1 (vorinostat 200 mg). Phase I protocol closed prematurely with no additional subjects enrolled. No analysis due to premature closure.
Groups:
- Phase I Dose Escalation of Vorinostat (200-400mg): Vorinostat 200 mg PO QD D1-14; Carbo 6 (AUC) D3; Etoposide 100 mg/m2 D1,2,3 Vorinostat, Carboplatin, Etoposide, SAHA
  Vorinostat, Carboplatin, Etoposide: Sequential cohorts of 3-6 patients will be entered to the following dose levels: Level 1 - Days 1-14: Vorinostat 200 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Level 2 - Days 1-14: Vorinostat 300 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2; Level 3: Days 1-14: Vorinostat 400 mg po QD; Day 3: Carboplatin 6 AUC; Days 1,2,3: Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each patient.
Arm/Group | Phase I Dose Escalation of Vorinostat (200-400mg)
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate Overall Survival of Patients With Extensive Disease SCLC Receiving Carboplatin, Etoposide, and a Fixed Dose (300mg) of Vorinostat
Description: For the purpose of this study, overall survival is defined as the percentage of participants who are alive at two years post initiation of study treatment.
Time Frame: 2 years, not analyzed
Population: One participant enrolled on Phase II. Off treatment and off study prematurely due to concurrent health disorders.
Groups:
- Phase II Vorinostat 300mg With Carboplatin and Etoposide: Participants with extensive disease SCLC receiving carboplatin, Etoposide, and a fixed dose (300mg) of vorinostat.
  Days 1-4 Vorinostat 300mg po QD; Day 3 Carboplatin 6 AUC; Days 1,2,3 Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each participant.
Arm/Group | Phase II Vorinostat 300mg With Carboplatin and Etoposide
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluate Objective Response Rate Among Patients With Extensive Disease SCLC Receiving Carboplatin and Etoposide With a Fixed Dose of Vorinostat.
Description: Eligibility limits the study population to those who have measurable disease pre-treatment. This secondary outcome measure was intended to objectively evaluate disease response and survival rate in recipients of the investigational medication regimen. Disease response was performed using standard diagnostic imaging. Tumor markers and cytology may be used to support the imaging results. Objective response rate was defined as progression-free survival (PFS) among treatment recipients. PFS, is defined as time (in months) from entry to clinical evidence of disease progression or death without progression. The clinical trial closed prematurely due to low accrual. For this reason, an analysis of this secondary objective would not be meaningful. No analysis done.
Time Frame: 2 years, not analyzed
Population: One participant enrolled and treated in the Phase II portion. Participant rendered off treatment and off study prior to completion due to concurrent health disorders. The clinical trial closed prematurely due to low accrual. For this reason, an analysis of this secondary objective would not be meaningful. No analysis done.
Groups:
- Phase II Vorinostat 300mg With Carboplatin and Etoposide: Participants with extensive disease small cell lung cancer who receive carboplatin plus etoposide with a fixed dose of vorinostat. Participants will receive: Days 1-4 Vorinostat recommended phase II dose po QD; Day 3 Carboplatin 6 AUC; Days 1,2,3 Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each participant.
Arm/Group | Phase II Vorinostat 300mg With Carboplatin and Etoposide
Number analyzed (Participants) | 0

4. Secondary Outcome: To Assess the Safety Profile and Define the Toxicities of Using a Fixed Dose (300mg) of Vorinostat With Carboplatin and Etoposide
Description: Evaluation of resultant adverse events that occurred with participants with extensive disease SCLC after initiating treatment using a fixed dose of vorinostat in combination with carboplatin and etoposide.
Time Frame: 2 years, not analyzed
Population: One participant enrolled in the Phase II portion and discontinued treatment prematurely due to concurrent health issues and hospitalization. No unanticipated adverse events occurred while on study. The study closed prematurely due to low accrual. No analysis conducted.
Groups:
- Phase II Vorinostat 300mg With Carboplatin and Etoposide: Participants with extensive disease SCLC receiving carboplatin, Etoposide, and a fixed dose (300mg) of vorinostat. Participants will receive on Days 1-4 Vorinostat 300mg po QD; Day 3 Carboplatin 6 AUC; Days 1,2,3 Etoposide 100 mg/m2. Treatment cycles will be repeated every 3 weeks. A maximum of 4 cycles will be administered to each participant.
Arm/Group | Phase II Vorinostat 300mg With Carboplatin and Etoposide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The time period for adverse event collection is from the time of consent to 30 days after last treatment cycle.
Description: Per clinicaltrials.gov standard definitions
Groups:
- Phase II: Vorinostat 300mg With Carboplatin and Etoposide: Phase 2 objective is to determine progression free survival among patients with extensive disease SCLC receiving carboplatin plus etoposide using an established dose of Vorinostat.
  Participants in Phase II received a "cycle" consisting of the NCI recommended Vorinostat dose with Carboplatin 6 AUC and Etoposide 100 mg/m2. Treatment cycles were repeated every 3 weeks. A maximum of 4 cycles were administered. A total of 35 participants were required for Phase II analysis. The Phase II study closed prematurely due to low accrual. Analysis of the primary and secondary objectives was not possible due to inadequate sample size.
- Phase I: Determine MTD Vorinostat (200mg-400mg): The original purpose of the Phase I portion was to establish the MTD of Vorinostat when provided with other chemotherapy (Carboplatin and Etoposide). Initial dose at 200mg, then 300, to a max of 400 mg. The first cohort at 200 mg did well with no dose limiting toxicities. After the enrollment of the 1st participant into cohort 2, the Phase I study was prematurely closed as concurrent NCI publications had established appropriate dose levels. The phase I portion was closed after the first 3 participants. Analysis of the objectives is not applicable due to premature closing.
Arm/Group | Phase II: Vorinostat 300mg With Carboplatin and Etoposide | Phase I: Determine MTD Vorinostat (200mg-400mg)
All-Cause Mortality (participants affected / at risk) | 1/1 | 3/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: Vorinostat 300mg With Carboplatin and Etoposide (N=1) | Phase I: Determine MTD Vorinostat (200mg-400mg) (N=3)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) — Phlebitis (including superficial thrombosis); Hospitalization for Thrombophlebitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: Vorinostat 300mg With Carboplatin and Etoposide (N=1) | Phase I: Determine MTD Vorinostat (200mg-400mg) (N=3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (10) — Leukocytes (total WBC)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (11) — Neutrophils/granulocytes (ANC/AGC)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (10) — Platelets, low
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (5) — Nausea
Fatigue (General disorders) | 0 (0) | 3 (9) — Fatigue (asthenia, lethargy, malaise)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) — Hemoglobin, Low
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) — Glucose, serum-high (hyperglycemia)
Facial flushing (General disorders) | 0 (0) | 1 (3) — Flushing
Alkaline phosphatase, elevated (Metabolism and nutrition disorders) | 0 (0) | 3 (3) — Alkaline phosphatase
Insomnia (General disorders) | 0 (0) | 2 (4) — Insomnia
Vaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (3) — Infection with unknown ANC, vaginal
Alanine aminotransferase (ALT) elevation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — ALT, SGPT (serum glutamic pyruvic transaminase)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Decreased appetite
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1) — Bilirubin (hyperbilirubinemia)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Calcium, serum-low (hypocalcemia)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Productive cough
Erythema, skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Erythema to lips and leg patch
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) — Dry mouth/salivary gland (xerostomia)
Fever without neutropenia (General disorders) | 0 (0) | 1 (1) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — Hiccoughs (hiccups, singultus)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Infection with unknown ANC - Skin - cellulitis
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Magnesium, serum-high (hypermagnesemia)
Restlessness with irritibility (Nervous system disorders) | 0 (0) | 1 (1) — Mood alteration - Agitation
Anxiety (Nervous system disorders) | 0 (0) | 1 (1) — Mood alteration - anxiety
Abnormal dreams (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Nervous system disorders) | 0 (0) | 1 (2)
Pain, extremity/limb (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Pain - Throat/pharynx/larynx (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Potassium, serum-low (hypokalemia)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) — Sodium, serum-low (hyponatremia)
Ulceration, vaginal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Vaginal ulceration lesion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No